CLINICAL TRIAL: NCT06875947
Title: EFFECTS of MORINGA OLEIFERA LEAF MICRONIZED POWDERS on HEMATOLOGICAL PROFILES, PERIPHERAL BLOOD SMEAR, HEPCIDIN, AND CYTOKINES (IL-1 DAN IL-6) OF PREGNANT WOMEN WITH IRON DEFICIENCY ANAEMIA
Brief Title: EFFECTS of MORINGA OLEIFERA LEAF POWDERS on HEMATOLOGICAL PROFILES IN PREGNANT WOMEN WITH IRON DEFICIENCY ANAEMIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, H. Awie Darwizar, M.D., Sp.OG., D.MAS., MMRS., FIHFAA, Principal Investigator, Department of Obstetrics and Gynecology, Fakultas Kedokteran Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 159/UN.6.KEP/EC/2025
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Iron Deficiency Anemia of Pregnancy; Pregnancy Complications; Inflammation; Moringa Oleifera; Cytokines (IL-1, IL-6); Hepcidin
Keywords: Iron Deficiency Anemia; Pregnancy Complications, Hematologic; Moringa oleifera; Dietary Supplements; Hepcidins; Interleukin-1; Interleukin-6; Erythrocyte Indices; Randomized Controlled Trial; Pregnancy; Nutritional Therapy; Oxidative Stress; Traditional Medicine; Phytotherapy
MeSH Terms: conditions — Pregnancy Complications; Inflammation; Anemia, Iron-Deficiency; Pregnancy Complications, Hematologic | interventions — Capsules; Folic Acid

STUDY DESIGN:
Intervention Model Description: This clinical study uses a Parallel Assignment Model, where participants are randomly allocated into two independent groups. Group A (Intervention) will receive Moringa Oleifera Leaf Micronized Powders (MOLMP) capsules combined with standard iron tablets, while Group B (Control) will receive standard iron tablets alone. Both groups will be followed simultaneously over a 60-day intervention period, with regular monitoring of hematological parameters, iron biomarkers, and inflammatory cytokines. This model allows direct comparison between the intervention and control groups to assess the efficacy and safety of Moringa Oleifera in improving iron deficiency anemia outcomes during pregnancy.
Masking Description: This study will be conducted without blinding, meaning that both the participants and researchers will be aware of the treatment assignments. This approach is chosen to facilitate close monitoring of adherence, safety, and any potential side effects during the intervention period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Moringa Oleifera Leaf Micronized Powders + Standard Iron Tablets (Experimental): Participants in this group will receive Moringa Oleifera Leaf Micronized Powders (MOLMP) 3×650 mg/day in capsule form, combined with standard iron tablets (Fe tablet 60 mg + Folic Acid 400 mcg/day) for 60 days.
  This intervention aims to evaluate the combined effect of Moringa Oleifera and standard iron supplements on hematological parameters, iron homeostasis, and inflammatory markers in pregnant women with iron deficiency anemia.
  Interventions: Dietary Supplement: Moringa Oleifera Leaf Micronized Powders in Capsule; Drug: Standard Iron Tablets (Fe + Folic Acid)
- Active Comparator: Control Group - Standard Iron Tablets Only (Active Comparator): Participants in this group will receive only standard iron tablets (Fe tablet 60 mg + Folic Acid 400 mcg/day) for 60 days.
  This arm serves as the control group to compare the effectiveness of standard iron therapy alone versus the combined intervention (MOLMP + Iron Tablets).
  Interventions: Drug: Standard Iron Tablets (Fe + Folic Acid)

INTERVENTIONS:
Dietary Supplement: Moringa Oleifera Leaf Micronized Powders in Capsule — Moringa Oleifera Leaf Micronized Powders (MOLMP)
  Source: Derived from finely ground Moringa Oleifera leaves using micronization technology to enhance bioavailability.
  Dosage: 650 mg per capsule, taken three times daily (1,950 mg/day). Administration Duration: 60 days. Monitoring: Self-administration under weekly compliance checks.
  Other Names: Bubuk Halus Daun Kelor
  Arms: Intervention Group - Moringa Oleifera Leaf Micronized Powders + Standard Iron Tablets
Drug: Standard Iron Tablets (Fe + Folic Acid) — Dosage: One tablet containing 60 mg iron and 400 mcg folic acid per day. Administration Duration: 60 days.
  Other Names: Tablet Tambah Darah

SUMMARY:
Title: The Effect of Moringa Oleifera Leaf Micronized Powders on Hematological Profile, Hepcidin, and Cytokines (IL-1 and IL-6) in Pregnant Women with Iron Deficiency Anemia

Study Description:

Iron deficiency anemia is one of the most common health problems affecting pregnant women worldwide, especially in developing countries like Indonesia. This condition can cause serious complications for both mothers and babies, such as premature birth, low birth weight, and increased risk of maternal mortality. Despite the availability of iron supplements as a standard treatment, many women experience side effects such as nausea, constipation, and poor absorption, which often lead to low adherence to the medication.

This clinical study aims to explore the potential of Moringa Oleifera leaf micronized powders (finely ground Moringa leaf powder) as a natural, plant-based supplement to help improve hemoglobin levels in pregnant women suffering from iron deficiency anemia. Moringa leaves are known for their rich nutritional content, including iron, antioxidants, and anti-inflammatory compounds, making them a promising alternative to traditional iron supplements.

The study will involve 72 pregnant women between 28-32 weeks of gestation diagnosed with iron deficiency anemia. Participants will be randomly assigned into two groups:

Group A will receive Moringa leaf capsules along with standard iron tablets. Group B will receive only standard iron tablets as the control group. The intervention will last for 60 days, during which participants will undergo regular blood tests to measure hemoglobin levels, iron status markers (hepcidin, TIBC), and inflammatory cytokines (IL-1 and IL-6). The study will also monitor the safety of Moringa leaf supplements, including liver and kidney functions.

Hypothesis: The study hypothesizes that adding Moringa Oleifera leaf micronized powders to standard iron therapy will significantly improve hemoglobin levels, iron status, and reduce inflammation in pregnant women with iron deficiency anemia compared to iron tablets alone.

This research is expected to provide scientific evidence supporting the use of Moringa leaves as a safe, effective, and affordable alternative therapy to help combat iron deficiency anemia during pregnancy.

DETAILED DESCRIPTION:
Title: The Effect of Moringa Oleifera Leaf Micronized Powders on Hematological Profile, Hepcidin, and Cytokines (IL-1 and IL-6) in Pregnant Women with Iron Deficiency Anemia

Background and Rationale:Iron deficiency anemia (IDA) remains a significant public health challenge during pregnancy, especially in low-to-middle-income countries. The condition affects both maternal and fetal health, increasing the risk of preterm delivery, low birth weight, and maternal mortality. Despite the widespread use of conventional iron supplements, the prevalence of anemia in pregnant women in Indonesia consistently exceeds 40% over the last two decades (WHO, 2022). Conventional iron tablets often result in gastrointestinal side effects, poor adherence, and limited bioavailability, highlighting the urgent need for alternative therapies.

Moringa Oleifera leaves have been widely recognized for their high nutritional value, containing essential micronutrients such as iron, calcium, vitamin C, and antioxidants. Emerging studies suggest that Moringa leaves have hematopoietic, anti-inflammatory, and antioxidant properties, making them a promising adjunctive therapy for iron deficiency anemia. However, high-quality clinical trials evaluating their efficacy and safety in pregnant women are still limited.

This randomized controlled trial (RCT) will investigate whether Moringa Oleifera Leaf Micronized Powders (MOLMP) combined with standard iron supplementation improves hematological parameters and reduces inflammation compared to iron supplementation alone in pregnant women with IDA.

Study Design:

Type: Open-labeled, randomized controlled trial (RCT) Allocation: 1:1 Randomized Allocation Intervention Model: Parallel Groups Masking: None (Open Label) Study Duration: 60 Days Sample Size: 72 participants (36 in each group) Study Site: Community Health Centers (Puskesmas Muka, Joglo, Cijedil, Karang Tengah) in Cianjur, West Java, Indonesia

Intervention Groups:

Group A (Intervention): Moringa Oleifera Leaf Micronized Powders (MOLMP) capsules (3x650 mg/day) + standard iron tablets (Fe tablet 60 mg + Folic Acid 400 mcg/day) Group B (Control): Standard iron tablets (Fe tablet 60 mg + Folic Acid 400 mcg/day) only

The Moringa Oleifera powder will be processed through micronization technology to increase bioavailability and optimize nutrient absorption.

Primary Outcome Measures:

Hemoglobin (Hb) levels Hematocrit (Hct) levels Erythrocyte Indices (MCV, MCH, MCHC) Serum Hepcidin levels (as a biomarker of iron homeostasis) Serum IL-6 (Pro-inflammatory cytokines)

Secondary Outcome Measures:

Serum IL-1β (Pro-inflammatory cytokines) Peripheral Blood Smear Analysis Total Iron Binding Capacity (TIBC) Reticulocyte Hemoglobin Content (RET-He) Red Cell Distribution Width (RDW-SD, RDW-CV) Liver Function Tests (SGOT, SGPT) Kidney Function Tests (Creatinine levels)

Methodology:

Participants will undergo screening and baseline laboratory tests on Day 0, followed by random allocation into two groups. All participants will receive standard antenatal care. Intervention products will be administered daily under self-administration supervision for 60 days. Compliance will be monitored through weekly visits, phone reminders, and supplement consumption diaries.

Blood samples will be collected at baseline (Day 0), and Day 60 to assess hematological parameters, iron status markers, and inflammatory biomarkers. Safety assessments will be conducted throughout the study to monitor liver and kidney function.

Randomization and Allocation Concealment:

Random allocation will be conducted using computer-generated random numbers. Participants will be assigned to either Group A or Group B with a 1:1 ratio.

Statistical Analysis Plan:

Baseline characteristics will be compared using Chi-square tests for categorical variables and Independent t-tests or Mann-Whitney U tests for continuous variables.

Primary outcomes will be analyzed using Repeated Measures ANOVA or Mixed Effects Models to evaluate changes over time.

Secondary outcomes will be analyzed using ANCOVA adjusted for baseline values and potential confounders.

Statistical significance will be set at p < 0.05.

Ethical Considerations:

The study has received ethical approval from the Ethics Committee of Universitas Padjadjaran (No: 159/UN6.KEP/EC/2025). Written informed consent will be obtained from all participants prior to enrolment. All procedures will comply with ICH-GCP (Good Clinical Practice) guidelines and the Declaration of Helsinki.

Risk and Safety Monitoring:

Potential side effects of Moringa Oleifera supplements include hypotension and hypoglycemia. Adverse events will be recorded using standardized Adverse Event Report Forms. Liver and kidney function will be closely monitored.

Data Confidentiality:

Participant data will be anonymized using unique identification codes. All information will be stored in encrypted databases and retained for a minimum of 10 years.

Expected Outcomes:

It is anticipated that the addition of Moringa Oleifera Leaf Micronized Powders will result in:

A significant increase in hemoglobin levels Improved iron homeostasis through reduced hepcidin levels Lower levels of pro-inflammatory cytokines (IL-1 and IL-6) Minimal side effects compared to standard iron tablets

Significance of Study:

If proven effective, Moringa Oleifera leaf powder could serve as a safe, natural, and cost-effective alternative to improve iron deficiency anemia in pregnant women, especially in resource-limited settings.

Due to an extension of the participant recruitment period, the anticipated timelines of the study have been updated. Participant recruitment is expected to continue until January 2026. The primary completion date defined as the date when the final participant receives the intervention and primary outcome data are collected, is anticipated to be March 2026. Final data collection for all study outcomes is anticipated to be completed by April 2026.

Principal Investigator:

H. Awie Darwizar, M.D., Sp.OG., D.MAS., MMRS., FIHFAA Email: adarwizar1512@gmail.com Phone: +62 812 2323 132

ELIGIBILITY:
Inclusion Criteria

1. Demographic Characteristics:

   * Women aged 18-44 years
   * Married, have a husband and/or family
   * Have an ID card
2. Clinical Characteristics:

   * Pregnant with a gestational age of 28 to <32 weeks
   * Live single fetus
   * Hemoglobin (Hb) 7 - < 11 g/dl
   * No congenital abnormalities
   * No complication (DM, infection, genetic disease) based on history taking, clinical signs and symptoms and treatment history.
   * Parity < 4
3. Geographical/Administrative Characteristics:

   * The study subjects (pregnant women) were located in the working area of the health facility where the study was conducted.

Health Facility where the study was conducted.

- Come to the health facility independently or by referral.

Exclusion Criteria:

* Pregnant women with high risk who dropped out or could not be followed up and pregnant women who gave birth prematurely.
* Allergy to Moringa Oleifera leaf micronized powders

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin Levels | Baseline (Day 0) and Day 60
  Measurement of hemoglobin concentration (g/dL) in venous blood to assess the improvement of anemia status in response to intervention. Hemoglobin is the primary indicator for anemia diagnosis and treatment effectiveness.
Hematocrit Levels | Baseline (Day 0) and Day 60
  Proportion of red blood cells to the total blood volume (%) to evaluate anemia severity and treatment response. Hematocrit indicates the volume percentage of red blood cells in blood samples.
Mean Corpuscular Volume (MCV) | Baseline (Day 0) and Day 60
  Measurement of the average size of red blood cells (fL) to classify anemia as microcytic, normocytic, or macrocytic, which reflects the effect of the intervention on red cell morphology.
Mean Corpuscular Hemoglobin (MCH) | Baseline (Day 0) and Day 60
  Measurement of the average concentration of hemoglobin in a given volume of red blood cells (g/dL), reflecting the effect of intervention on hemoglobin saturation within red blood cells.
Serum Hepcidin Levels | Baseline (Day 0) and Day 60
  Quantification of serum hepcidin (ng/mL) as a biomarker of iron homeostasis and iron absorption regulation. Hepcidin levels will help assess the intervention's role in modulating iron metabolism.
Serum IL-6 Levels | Baseline (Day 0) and Day 60
  Measurement of interleukin-6 (IL-6) concentration (pg/mL) in venous blood to evaluate the intervention's effect on systemic inflammation, which plays a critical role in iron metabolism.
Mean Corpuscular Hemoglobin Concentration (MCHC) | Baseline (Day 0) and Day 60
  Measurement of the average concentration of hemoglobin in a given volume of red blood cells (g/dL). MCHC reflects the hemoglobin saturation within erythrocytes and is used to assess the severity and type of anemia. Changes in MCHC indicate improvements in iron availability and erythropoiesis in response to supplementation.
Serum Iron | Baseline (Day 0) and Day 60
  Serum Iron represents the actual circulating iron available for erythropoiesis (red blood cell production). In IDA, serum iron levels decrease significantly due to depleted iron stores. Serum iron helps quantify the degree of iron deficiency and supports a more precise biochemical assessment of IDA when used alongside TIBC.

SECONDARY OUTCOMES:
Total Iron Binding Capacity (TIBC) | Baseline (Day 0) and Day 60
  Measurement of the blood's capacity to bind iron with transferrin (µg/dL), indicating iron availability and iron saturation.
Reticulocyte Hemoglobin Content (RET-He) | Baseline (Day 0) and Day 60
  Measurement of hemoglobin content in reticulocytes (pg), reflecting recent iron availability for erythropoiesis.
Red Cell Distribution Width - Standard Deviation (RDW-SD) | Baseline (Day 0) and Day 60
  Measurement of the variation in red blood cell size (fL), indicating anisocytosis related to iron deficiency anemia.
Red Cell Distribution Width - Coefficient of Variation (RDW-CV) | Baseline (Day 0) and Day 60
  Measurement of the coefficient of variation of red blood cell size distribution (%), providing additional information on anisocytosis severity.
Serum IL-1β Levels | Baseline (Day 0) and Day 60
  Measurement of serum interleukin-1 beta (IL-1β) concentration (pg/mL) to evaluate systemic inflammatory response.
Serum Glutamate Pyruvate Transaminase (SGPT) | Baseline (Day 0) and Day 60
  Measurement of SGPT levels (U/L) to assess liver function and monitor potential hepatotoxicity of the intervention.
Serum Glutamate Oxaloacetate Transaminase (SGOT) | Baseline (Day 0) and Day 60
  Measurement of SGOT levels (U/L) to evaluate liver function and detect potential hepatotoxicity of the intervention.
Serum Creatinine Levels | Baseline (Day 0) and Day 60
  Measurement of serum creatinine (mg/dL) to assess kidney function and monitor potential nephrotoxicity of the intervention.
Peripheral Blood Smear Analysis | Baseline (Day 0) and Day 60
  Microscopic evaluation of red blood cell morphology to detect changes such as hypochromia, microcytosis, anisocytosis, and poikilocytosis. This analysis provides supportive evidence for anemia classification and intervention effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusat Kesehatan Masyarakat (PUSKESMAS), Cianjur, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Plan Description :
  De-identified individual participant data (IPD) will be shared upon reasonable request for research purposes. The data will include:
  * Primary outcomes: Hemoglobin, hematocrit, erythrocyte indices, Hepcidin, IL-6
  * Secondary outcomes: Peripheral blood smear, iron metabolism markers ( TIBC), inflammatory markers (IL-1)
  * Additional parameters: RDW-SD, RDW-CV, Ret-He, SGOT, SGPT, creatinine Data will be stripped of all personal identifiers to ensure confidentiality and comply with ethical standards.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting documents will be available 6 months after publication of study results and will remain accessible for 5 years.
Access Criteria: Researchers affiliated with recognized academic or healthcare institutions may submit a formal request to access the data. Applications must be sent to the Principal Investigator at adarwizar1512@gmail.com. Requests will be reviewed to ensure compliance with ethical and scientific standards. Approved researchers must sign a Data Use Agreement (DUA). Data will be provided in anonymized format for scientific and academic purposes only.

REFERENCES:
- [Background] Pareek A, Pant M, Gupta MM, Kashania P, Ratan Y, Jain V, Pareek A, Chuturgoon AA. Moringa oleifera: An Updated Comprehensive Review of Its Pharmacological Activities, Ethnomedicinal, Phytopharmaceutical Formulation, Clinical, Phytochemical, and Toxicological Aspects. Int J Mol Sci. 2023 Jan 20;24(3):2098. doi: 10.3390/ijms24032098. PMID 36768420
- [Background] Stohs SJ, Hartman MJ. Review of the Safety and Efficacy of Moringa oleifera. Phytother Res. 2015 Jun;29(6):796-804. doi: 10.1002/ptr.5325. Epub 2015 Mar 24. PMID 25808883
- [Background] Weiss G, Ganz T, Goodnough LT. Anemia of inflammation. Blood. 2019 Jan 3;133(1):40-50. doi: 10.1182/blood-2018-06-856500. Epub 2018 Nov 6. PMID 30401705
- [Background] de Barros MC, Silva AGB, Souza TGDS, Chagas CA, Machado JCB, Ferreira MRA, Soares LAL, Xavier VL, de Araujo LCC, Borba EFO, da Silva TG, Alves RRV, Coelho LCBB, de Oliveira AM, Napoleao TH, Paiva PMG. Evaluation of acute toxicity, 28-day repeated dose toxicity, and genotoxicity of Moringa oleifera leaves infusion and powder. J Ethnopharmacol. 2022 Oct 5;296:115504. doi: 10.1016/j.jep.2022.115504. Epub 2022 Jun 26. PMID 35760258
- [Background] Vyoral D, Jiri Petrak. Therapeutic potential of hepcidin - the master regulator of iron metabolism. Pharmacol Res. 2017 Jan;115:242-254. doi: 10.1016/j.phrs.2016.11.010. Epub 2016 Nov 17. PMID 27867027